CLINICAL TRIAL: NCT03997422
Title: Hepatic Energy Fluxes, NASH, and Vertical Sleeve Gastrectomy
Brief Title: Hepatic Energy Fluxes in NASH and NAS Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURG-2019-27704
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; NAS; Overweight or Obesity; Weight Loss; Bariatric Surgery Candidate
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vertical Sleeve Gastrectomy (VSG) (Experimental): Bariatric surgical procedure
  Interventions: Procedure: Vertical Sleeve Gastrectomy (VSG)

INTERVENTIONS:
Procedure: Vertical Sleeve Gastrectomy (VSG) — Vertical Sleeve gastrectomy will be performed using five laparoscopic ports using a 40 French Bougie as a template. If a hiatal hernia is identified it will be repaired. This practice has greatly reduced postoperative reflux disease (see human subjects protection). As VSG for patients with a BMI 30.0-34.9 kg/m2 is not covered by insurance the University hospital will cover costs for up to 24 patients.

SUMMARY:
Diseases along the nonalcoholic fatty liver disease spectrum, which are tightly coupled to the obesity epidemic, are soon to become the commonest indication for liver transplantation in the United States. Bariatric surgery shows great promise in the treatment of these diseases. The studies proposed herein will be the first to measure in humans the relationships among (i) the liver's ability to burn fat and make glucose, two of its primary functions; (ii) the severity of nonalcoholic fatty liver disease; and (iii) the responses to bariatric surgery. These experiments will support deeper future mechanistic investigations of the metabolic mechanisms underlying nonalcoholic steatohepatitis (NASH) improvement with bariatric surgery.

The premise of this study is that deranged hepatic mitochondrial metabolism is a key biomarker and mediator of the nonalcoholic fatty liver disease (NAFLD)/NASH continuum, and the central hypothesis the investigators will test is that preoperative hepatic fat oxidation and glucose production flux parameters differ between low versus high NAFLD activity score (NAS), and response of the liver to bariatric surgery can be predicted by preoperative fluxes.

DETAILED DESCRIPTION:
Twenty-five percent of the United States population has nonalcoholic fatty liver disease (NAFLD), a disease that includes hepatic fatty infiltration alone (simple steatosis) or steatosis plus inflammation, liver cell injury and death (nonalcoholic steatohepatitis [NASH]). NAFLD involving hepatic steatosis alone can be a stable clinical condition existing as the hepatic manifestation of insulin resistance. NASH develops in 25% of patients with NAFLD, and likely has additional pathologic underpinnings compared to steatosis alone. NASH leads to liver fibrosis, an elevated risk of cirrhosis and hepatocellular carcinoma and is likely to be the leading cause of liver transplantation in the U.S. The gold standard to distinguish probable uncomplicated NAFLD from NASH can be made using the histopathological nonalcoholic fatty liver disease score (NAS) score in which the sum of the categorical severity of steatosis, inflammation, and hepatocyte ballooning injury is ≥ 4, i.e., suggestive of NASH. Patients with obesity (BMI³30 kg/m2), type 2 diabetes (T2DM), age older than 45 years, and certain ethnicities are at high risk for developing NASH. In the U.S., the cost of management of NASH and its complications is $32 billion annually. Durable therapies are lacking for the NASH spectrum and an acceptable pharmaceutical intervention is not approved. Weight loss, achieved through lifestyle modification, is the cornerstone of therapy. Improvements in NAS are proportional to weight loss but weight loss does not reliably surpass 10% with lifestyle modification. Weight loss surgery (bariatric surgery) achieves dramatic weight loss. The vertical sleeve gastrectomy (VSG), a bariatric surgical procedure, can dramatically reduce (NAS) and favor NASH remission. Importantly, not all patients with NASH demonstrate histologic improvements following bariatric surgery, and in a small percentage of patients the disease may progress. Presently, it is not known what mechanistic biomarkers might prioritize steatosis, inflammation, or hepatocyte ballooning injury, and furthermore there are no known antecedent biomarkers of outcome of NAFLD with bariatric surgery. As the primary host for glucose and fat metabolism, the liver forms the critical nexus for whole body metabolism. In the setting of insulin resistance and NAFLD, glucose production becomes less responsive to the suppressive effects of insulin while de novo fat synthesis is enhanced in a paradoxical setting in which fat oxidation is not decreased. Mitochondrial b-oxidation of fatty acids normally produces acetyl-CoA which is terminally oxidized via the tricarboxylic acid (TCA) cycle, producing reducing equivalents needed for gluconeogenesis. While measured in uncomplicated human NAFLD, hepatic energy fluxes have never been formally measured in human NASH, and thus there is an unmet need to determine whether mitochondrial metabolism drives and/or predicts NAFLD progression/resolution, potentially yielding quantifiable predictive value over NAS alone. The research group has developed magnetic resonance spectroscopy (MRS)- based methods for quantifying hepatic oxidative energy fluxes and glucose metabolism ('hepatic energy fluxes') using administered dual 2H and 13C isotope tracers non-invasively and without imaging, requiring only collections of peripheral venous blood. These flux measurements will be performed at baseline in obese patients (BMI of 30-39.9 kg/m2) prior to VSG, who have all received preoperative liver biopsies for histopathological determination of NAS score, liver MRI-derived proton density fat fraction (PDFF) and elastography (MRE) assessment of fibrosis, and intravenous glucose tolerance tests (IVGTT) as a crude measure of insulin resistance. Then it will be determined how preoperative energy flux indices correlate with pre- and post-operative NAS, PDFF, and MRE indices. Thus, the premise of this study is that deranged hepatic mitochondrial metabolism is a key biomarker and mediator of the NAFLD/NASH continuum, and the central hypothesis the investigators will test is that preoperative hepatic fat oxidation and glucose production flux parameters differ between low versus high NAS, and response of the liver to bariatric surgery can be predicted by preoperative fluxes. It is anticipated that these preliminary observations will serve as proof-of-concept datasets supporting future R01 funding that comprehensively determine the role of hepatic oxidative fluxes in human NASH evolution and response to bariatric surgery. This will be first study to quantify hepatic metabolic fluxes in obese (BMI 30-39.9 kg/m2) adult patients with biopsy-proven NASH compared to NAFLD without NASH. This will also be the first study to correlate these findings to histopathological, radiographic, and clinical outcomes following VSG. Central parameters of hepatic energy fluxes, and the relative contributions of the liver's three carbon sources to endogenous glucose production (i.e., from PEP, glycogen, or glycerol), have not been quantified for in human NASH. Contributions of these metabolic indices preoperatively to VSG outcomes have not been interrogated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 67 years at eligible visit
* Diagnosed with NASH with a total NAS ≥ 3 including a ballooning score of at least 1, or non-NASH/NAFLD with a total NAS ≤3, or Diagnosed with T2DM or prediabetes, HbA1c< 8% , or CAP score greater than or equal to 248 on Fibroscan
* Body Mass Index (BMI) 30.0-55.0 kg/m2 at eligibility visit
* Willingness to accept surgical intervention after an individual seminar session
* All patients must have insurance with no exclusion for obesity related treatments or management of obesity surgery complications. This applies to all patients enrolled in the study
* Expect to live or work within approximately three-hour traveling time from the study clinic for the duration of the one-year trial
* Willingness to comply with the follow-up protocol and successful completion of the run-in
* Written informed consent
* Suitable for liver biopsy using the percutaneous approach
* Vulnerable populations will not be targeted for inclusion, but those noted in section 9.1 may be allowed to participate provided they met all of the inclusion and none of the exclusion criteria.

Exclusion Criteria:

* Cardiovascular event (myocardial infarction, acute coronary syndrome, coronary artery angioplasty or bypass, stroke) in the past six months.
* Current evidence of congestive heart failure, angina pectoris, or symptomatic peripheral vascular disease.
* Cardiac stress test indicating that surgery or IMM would not be safe.
* Pulmonary embolus or thrombophlebitis in the past six months
* Cancer of any kind (except basal cell skin cancer or cancer in situ) unless documented to be disease-free for five years.
* Significant anemia (hemoglobin 1.0 g/dL or more below normal range) or history of coagulopathy.
* Serum creatinine >1.5 mg/dL.
* Serum total bilirubin greater than the upper limit of normal in the absence of Gilbert's syndrome, or alkaline phosphatase or ALT or AST greater than 2.5 the upper limit of normal. Elevated INR.
* Alcohol intake more than one drink or >20 grams per day
* History of stomach surgery, bile duct surgery, pancreatic surgery, splenectomy, or colon resection.
* Gastric or duodenal ulcer in the past six months.
* History of intra-abdominal sepsis (except for uncomplicated appendicitis or diverticulitis more than six months prior to enrollment).
* Previous organ transplantation.
* Self-reported HIV-positive status, active tuberculosis, active malaria, chronic hepatitis B or C, or cirrhosis
* Currently pregnant or nursing, or planning to become pregnant in the next two years.
* History of alcohol, drug, or opioid dependency (excluding nicotine) in the past five years.
* Active psychosocial or psychiatric problem that is likely to interfere with adherence to the protocol.
* Depression A CESD score more than 17 and a psychologist determination that the patient is not a good fit for surgery.
* Presence of any chronic or debilitating disease that would make adherence to the protocol difficult.
* 12-lead EKG indicating that surgery would not be safe.
* Serum c-peptide <1.0 ng/ml post prandial.
* Exclusions may also be made at the discretion of the attending physician or the eligibility committee.
* Contraindication to MRI scanning. MRI contraindications are assessed by MR technologists on the day of scanning using a standard safety screening form.
* History of endoscopy demonstrating esophagitis or Barretts changes in the esophagus. Any history of dysphagia.
* Treatment with drugs associated with nonalcoholic fatty liver disease (amiodarone, methotrexate, oral glucocorticoids at doses greater than 5 mg/day, tamoxifen, estrogens at doses greater than those used for hormone replacement or contraception, anabolic steroids, valproic acid) for more than 4 weeks within the last 2 months prior to the initial screening.
* Treatment with pioglitazone or high-dose vitamin E (>400 IU/day) within the last 2 months prior to the initial screening.

Ages: 40 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic Energy Fluxes | 12 months
  Non-invasive dual isotope tracer-coupled magnetic resonance spectroscopy (MRS) will be used to measure tricarboxylic acid cycle (TCA) flux, anaplerosis, and gluconeogenesis.
  Outcome reported in micromols per minute per kg of lean body mass.

SECONDARY OUTCOMES:
Histologic improvements in NAFLD Activity Score (NAS) | 12 months
  The scale used is NAS - this is the NAFLD (Nonalcoholic Fatty Liver Disease) Activity Score.
  The NAS was developed to provide a numerical score for patients who most likely have NASH. Accordingly, NAS is the sum of the separate scores for steatosis (0-3), hepatocellular ballooning (0-2) and lobular inflammation (0-3). NAS scores of 0-2 are largely considered not diagnostic of NASH, scores of 3-4 are often considered not diagnostic, borderline, or potentially positive for NASH. Scores of 5-8 are largely considered diagnostic of NASH.
  It is expected that the addition of VSG to lifestyle modification will result in more robust histologic improvements in NAFLD Activity Score (NAS) compared to lifestyle modification alone.

CONTACTS AND LOCATIONS:
Overall Officials: Sayeed Ikramuddin, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No